CLINICAL TRIAL: NCT01261754
Title: A Phase I Study of the PK, Tissue Distribution and Metabolism of Small Molecule Inhibitors of Prostate Specific Membrane Antigen, 99mTc-MIP-1404 and 99mTc-MIP-1405, in Patients With Metastatic Prostate Adenocarcinoma and Healthy Volunteers
Brief Title: A Study of 99mTc-MIP-1404 and 99mTc-MIP-1405 in Patients With Metastatic Prostate Adenocarcinoma and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: TcTx-P101
Record Dates: First submitted 2010-11-18; First posted 2010-12-16 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
Keywords: Metastatic Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — technetium 99m 1-(1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)-2-((1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)methyl)-9,14-dioxo-2,8,13,15-tetraazaoctadecane-7,12,16,18-tetracarboxylic acid); technetium 99m 7-amino-1-(1-(carboxymethyl)-1H-imidazol-2-yl)-2-((1-(carboxymethyl)-1H-imidazol-2-yl)methyl)-8,16-dioxo-2,9,15,17-tetraazaicosane-14,18,20-tricarboxylic acid)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metastatic prostate adenocarcinoma (Active Comparator)
  Interventions: Radiation: 99mTc MIP 1404; Radiation: 99mTc MIP 1405
- Healthy Volunteers (Active Comparator)
  Interventions: Radiation: 99mTc MIP 1404; Radiation: 99mTc MIP 1405
- Newly Diagnosed, High-Risk Prosate Cancer Patients (Active Comparator)
  Interventions: Radiation: 99mTc MIP 1404; Radiation: 99mTc MIP 1405

INTERVENTIONS:
Radiation: 99mTc MIP 1404 — Subjects will be administered a single 20 (± 3) mCi intravenous (IV) injection of 99mTc MIP 1404
Radiation: 99mTc MIP 1405 — Subjects will be administered a single 20 (± 3) mCi intravenous (IV) injection of 99mTc MIP 1405

SUMMARY:
This is a single-blind, randomized, cross-over design. Patients with metastatic prostate adenocarcinoma; newly diagnosed, high-risk patients with prostate adenocarcinoma; and healthy subjects will be administered a single intravenous dose of each of the study drugs 99mTc MIP 1404 and 99mTc MIP 1405 administered approximately 14 to 21 days apart.

DETAILED DESCRIPTION:
This trial is a single-blind, randomized, cross-over design. Up to six patients with confirmed metastatic prostate adenocarcinoma; six newly diagnosed, high-risk patients with prostate adenocarcinoma; and up to six healthy volunteers will receive 20.0 (± 3) mCi of intravenously administered 99mTc MIP 1404 or 99mTc MIP 1405. Whole-body planar scintigraphic images will be acquired at various times post-injection over 24 hours. A pelvic SPECT/CT image will be acquired on the first day. Blood and urine will be collected for pharmacokinetic measurements and metabolic analysis over 24 hours. Each patient will receive an initial study drug administration and a second study drug administration approximately 14 to 21 days after the first. A final follow-up visit will occur approximately 2-3 weeks after the second study drug.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be enrolled in this study.

1. Male aged 21 years or older.
2. Ability to provide signed informed consent and willingness to comply with protocol requirements.
3. Participants must agree to use condoms for a period of seven days after each injection, if engaged in sexual activity.

Additional Inclusion Criteria for Patients:

i. Histologic diagnosis of prostate cancer by validated medical history. (Pathology report, if available).

ii. Evidence of metastatic disease demonstrated by a documented abnormal bone scan, CT scan, or MRI plus a Clinical Stage 3 and Gleason Score ≥ 8.

iii. Karnofsky performance is ≥ 60.

Additional Inclusion Criteria for Healthy Volunteers:

i. PSA laboratory assessment within normal range (PSA < 4 ng/ml). ii. Normal findings on a digital rectal examination. iii. Hemoglobin and hematocrit within normal range.

Exclusion Criteria:

Participants must NOT meet any of the following criteria to be enrolled in this study.

1. Received an investigational compound and/or medical device or is part of an investigational study within the past 30 days before enrollment into this study.
2. Subject was administered a radioisotope within 5 physical half lives of that radioisotope prior to study enrollment
3. Have any medical condition or other circumstances which, in the opinion of the Investigator, would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post dose follow-up examinations.
4. Participant is determined by the Investigator to be clinically unsuitable for the study.
5. Serum creatinine ≥ 2.0 mg/dl
6. Total bilirubin ≥ 2.0 mg/dl
7. Liver transaminases ≥ 1.5 x ULN
8. Platelet count < 150,000/mm3
9. Absolute neutrophil count (ANC) < 2,000/mm3.
10. Hematocrit < 30% or hemoglobin < 10 g/dl.
11. Abnormal coagulation profile (PT, PTT or INR) > 1.3 ULN unless on therapeutic anticoagulation.

Additional Exclusion Criteria for Patients:

Patients will be excluded from the study if any of the following criteria are observed:

i. Androgen deprivation therapy or other forms of hormonal therapy not stable for a period of 14 days prior to screening.

ii. Subject has received a permanent prostate brachytherapy implant within the last 3 months for 103Pd implants; or 12 months for 125I implants.

iii. Subject on or expected to be starting cytotoxic chemotherapy during the study period.

iv. Has had any other malignancies within the past year, other than basal or squamous cell carcinoma of the skin, diagnosis and location must be defined or be defined as clinically controlled or treated to complete response.

Additional Exclusion Criteria for Healthy Volunteers:

Healthy Volunteers will be excluded from the study if any of the following criteria are observed:

i. Have had any malignancies within 5 years other than basal or squamous cell carcinoma of the skin.

ii. History of known prostate adenocarcinoma, prostate surgery/biopsy, prostatitis and/or symptoms suggestive of or associated with possible prostatitis within 6 months of enrollment.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety of Administered dose | From the time of signed ICF through 2 weeks post injection of the second study drug administration (up to 8 weeks total for each subject)
  The safety data will be summarized for all patients receiving at least one dose of study drug. Summary tables, including change from pre dose to post dose where applicable, will be presented for the following safety endpoints:
  * Treatment emergent adverse events
  * Clinical Laboratory Evaluations
  * Physical examination, vital signs, and ECGs
Pharmacokinetics of Administered Dose | From the time of signed ICF through 2 weeks post injection of the second study drug administration (up to 8 weeks total for each subject)
  Standard PK parameters of 99mTc-MIP-1404 and 99mTc-MIP-1405 will be calculated, including but not limited to: clearance, distribution half-life, elimination half-life, mean residence time and maximum concentration. These PK parameters will be listed by subject and summarized. Blood clearance and urinary recovery over time will be displayed in figures. Urine metabolites and impurities of 99mTc-MIP-1404 and 99mTc-MIP-1405 will be listed by subject and summarized.
  The PK population will be used in the analysis of pharmacokinetics and metabolism.
Biodistribution of Administered Dose | : From the time of signed ICF through 2 weeks post injection of the second study drug administration (up to 8 weeks total for each subject)
  Percent of injected activity (%IA) in a set of source organs will be determined by comparing a reference whole body scan to subsequent whole body scans to determine percentage of administered activity for source organs at the various scanning times. This biodistribution data will then be used to mathematically model source organ residence times, which will be used to estimate radiation absorbed dose to target organs. Percent injected activity and estimated residence times will be summarized by organ.

SECONDARY OUTCOMES:
Excretion of administered dose | From the time of signed ICF through 2 weeks post injection of the second study drug administration (up to 8 weeks total for each subject)
  Standard PK parameters of 99mTc-MIP-1404 and 99mTc-MIP-1405 will be calculated, including but not limited to: clearance, distribution half-life, elimination half-life, mean residence time and maximum concentration. These PK parameters will be listed by subject and summarized. Blood clearance and urinary recovery over time will be displayed in figures. Urine metabolites and impurities of 99mTc-MIP-1404 and 99mTc-MIP-1405 will be listed by subject and summarized.
  The PK population will be used in the analysis of pharmacokinetics and metabolism.
Dosimetry of administered dose | From the time of signed ICF through 2 weeks post injection of the second study drug administration (up to 8 weeks total for each subject)
  To calculate the estimated radiation dosimetry to normal organs based on the pharmacokinetic and normal tissue distribution in patients with confirmed metastatic prostate adenocarcinoma and in healthy volunteers
Metabolism of administered dose | From the time of signed ICF through 2 weeks post injection of the second study drug administration (up to 8 weeks total for each subject)
  Standard PK parameters of 99mTc-MIP-1404 and 99mTc-MIP-1405 will be calculated, including but not limited to: clearance, distribution half-life, elimination half-life, mean residence time and maximum concentration. These PK parameters will be listed by subject and summarized. Blood clearance and urinary recovery over time will be displayed in figures. Urine metabolites and impurities of 99mTc-MIP-1404 and 99mTc-MIP-1405 will be listed by subject and summarized.
  The PK population will be used in the analysis of pharmacokinetics and metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J Goldsmith, MD, Principal Investigator — New York Presbyterian Hospital - Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital - Weill Medical College of Cornell University, New York, New York, United States